CLINICAL TRIAL: NCT07016256
Title: Effect of Different Oral Splints on the Maximum Bite Force in TMD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Vina del Mar (Other)
Responsible Party: Principal Investigator, Nicolás Pinto Pardo, Nicolas Pinto-Pardo, Universidad Vina del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UVMODO012025
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Muscular TMD
Keywords: TMD; oral splints; lucia jig; Sved splint; Occlusal splint; orofacial pain; muscular pain
MeSH Terms: conditions — Facial Pain; Myalgia

STUDY DESIGN:
Intervention Model Description: 75 men and 75 women diagnosed with muscular TMD, dividen in 3 groups (25 patients each) to evaluate 3 different oral splints on the maximum bite force
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lucia jig (Experimental): Lucia jig splint
  Interventions: Device: intraoral devices
- Sved splint (Experimental): Sved splint
  Interventions: Device: intraoral devices
- Occlusal splint (Experimental): Occlusal splint
  Interventions: Device: intraoral devices

INTERVENTIONS:
Device: intraoral devices — Intraoral devices not registed with a patent

SUMMARY:
The goal of this clinical trial is to evaluate whether three different types of intraoral splints can increase maximal voluntary mandibular clenching force in adults diagnosed with myogenous temporomandibular disorders (TMD). The main questions it aims to answer are:

Do intraoral splints enhance maximal clenching force in patients with muscle-related TMD? Is there a difference in the effectiveness of the three splint designs in improving muscle strength? Researchers will compare the effects of each splint within the same participants to determine which one most effectively increases clenching force.

Participants will:

Undergo baseline assessment of maximal mandibular clenching force Use each intraoral splint for a 30-day period Complete follow-up assessments after each intervention phase

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effect of three different types of intraoral splints on maximal voluntary bite force in patients diagnosed with myogenous temporomandibular disorders (TMD). A total of 150 participants were recruited, consisting of 75 men and 75 women. Each gender group was evenly divided into three intervention arms:

25 participants received the Lucia Jig splint 25 participants received the Sved splint 25 participants received the Occlusal splint All participants were previously diagnosed with muscle-related TMD by a qualified clinician. Each participant served as their own control. Baseline measurements of maximum bite force were recorded prior to the intervention using a gnatodynamometer (Kratos, Brazil). Measurements were taken in two anatomical zones: the incisal zone and the molar zone.

For each zone, three consecutive bite force measurements were recorded, with a 5-minute rest interval between each trial. The average of the three measurements was calculated and used as the baseline value for each zone.

Participants were instructed to use their assigned intraoral splint nightly for a period of 30 days. After this period, they returned for a follow-up assessment. The same measurement protocol was repeated: three bite force recordings in both the incisal and molar zones, each separated by a 5-minute interval. The average of these three post-intervention values was calculated for comparison with the baseline.

This within-subject design allows for the evaluation of changes in bite force attributable to each splint type, and for comparison across the three splint designs. The study seeks to determine whether intraoral splints can enhance muscle strength in patients with myogenous TMD, and which design is most effective in doing so.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with muscular TMD
* Not using ant
* Non pregnant women.
* Not under convulsive, chronic pain, antidepresive, antihypertensive, pharmacological treatments
* Without systemic pathologies.

Exclusion Criteria:

* Treatment for chronic pain, depression, hypertension, convulsion condition with or without medication.
* Regular use of benzodiazepines.
* Systemic pathologies
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Maximum bite force in the incisal and molar zones | From enrollment to 30 days after splint utilization
  Each patient will be tested at the beginning of the clinical trial on the maximum bite force in the incisal zone, and after 30 days post splint utilization

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Viña del Mar, Viña del Mar, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet really, so we need more time to consider that